CLINICAL TRIAL: NCT06392035
Title: Determining the Effect of Nutrition Education Based on PENDER's Health Promotion Model on the Breakfast Habits of Secondary School Students
Brief Title: Breakfast Training Based on PENDER's Health Promotion Model (HPM)
Acronym: (HPM)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Collaborators: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Secil Duran Yilmaz, Lecturer, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 13562490-299-55
Record Dates: First submitted 2024-04-16; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Health Education
Keywords: Breakfast Consumption; School Age Children; Health Promotion Model
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: In the research, an experiment and a control group will be selected.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention will be made to the participants in the control group. A pre-test will be administered before the study and a post-test will be administered after the study.
- Intervention Group (Experimental): Secondary schools located in Karaman city center will be visited. The researcher will introduce himself and explain the purpose of the research.
  A research inclusion form will be applied to those who agree to participate in the research.
  "Sociodemographic Data Form", "Nutrition Behavior Scale", "Parental Questionnaire" and "Tool for Measuring the Health Promotion Model Related to Breakfast Consumption" will be applied as pre-test forms to the participants who meet the inclusion criteria. Participants will be assigned randomization by someone other than the researcher. After randomization assignment, a 6-week web-based training based on PENDER's Health Promotion Model, prepared in line with the literature, will be applied.
  Interventions: Other: health education, web-based education

INTERVENTIONS:
Other: health education, web-based education — Data collection tools will be filled in by two study groups (experimental group, control group) and based on the pre-test results of both groups, Pender's SGM-based breakfast training will be given only to the experimental group. No intervention will be made to the control group. In this study, a total of 6 sessions will be held for the experimental group for 6 weeks (one session per week), each lasting 40 minutes. In these sessions, web-based training will be given every week according to the components of the model and will be supported with written and visual brochures.
  Arms: Intervention Group

SUMMARY:
Nutrition of school-age children is very important. Children at this age need to eat three main meals and at least one snack every day. Breakfast, among the main meals, is an important component of a healthy diet and is vital for healthy and normal development, especially in children and adolescents. T.R. According to TÜBER prepared by the Ministry of Health, the most frequently skipped meal among school-age children is breakfast. It is necessary to raise awareness in parents and children about regular breakfast consumption and frequency and to instill healthy lifestyle behaviors. It is aimed to regulate breakfast consumption and frequency in parents and children with a web-based training based on PENDER Health Promotion Model (HGM).

DETAILED DESCRIPTION:
Before starting the study, students and parents will be informed in writing and verbally. Then, a pre-test will be applied with the specified data collection tools to students and parents who agree to participate in the research. Then, a 6-week web-based training on breakfast consumption based on PENDER's Health Promotion Model will be given. After the training, a post-test will be applied with data collection tools. Then the pre-test and post-test data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* • Being a 7th grade student of secondary school,

  * Not having a chronic disease
  * Students who voluntarily agreed to participate in the research and received consent from their parents.

Exclusion Criteria:

* • Not being a 7th grade student of secondary school,

  * Having a chronic disease
  * Students who do not agree to participate in the research voluntarily and whose parents' consent cannot be obtained

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2024-05-22 (Estimated); Primary Completion 2024-07-22 (Estimated); Study Completion 2024-07-22 (Estimated)

PRIMARY OUTCOMES:
Teaching children the habit of regular breakfast | at the end of the 1th weeks
  Children will be taught regular breakfast habits. Here, weight, height and BMI status will be examined. Weight in kilograms; Height will be measured in metres. Weight and height will be combined. BMI will be reported in kg/m^2.
Teaching children the habit of regular breakfast | at the end of the 6th weeks
  Children will be taught regular breakfast habits. Here, weight, height and BMI status will be examined. Weight in kilograms; Height will be measured in metres. Weight and height will be combined. BMI will be reported in kg/m^2.

SECONDARY OUTCOMES:
"Health Promotion Model Related to Breakfast Consumption (first week) ) | at the end of the 1th weeks
  Health Promotion Model Related to Breakfast Consumption scale consists of 10 sub-dimensions and 58 items.
  Previous Relevant Behavior (first 10 questions - score range 10-50) Perceived Usefulness (questions 11-16 - score range 6-30) Perceived Obstacles (questions 17-24-score range 8-40) Perceived Self-Efficacy (questions 25-32 - score range 8-40) Positive Impact (33,34 questions - score range 2-10) Negative Impact (35,36 questions - score range 2-10) Interpersonal Influences (questions 37-46 - score range 10-50) Situational Effects (questions 47,48,49 - score range 3-15) Instant Competing Demands and Preferences (questions 50,51,52,53 - score range 4-20) Planning Commitment (questions 54-58 - score range 5-20)
Nutrition behavior scale (first week) | at the end of the 1th weeks
  Children's food consumption was evaluated with the "Nutrition Behavior Scale" developed within the scope of CATCH (Child and Adolescent Trial for Cardiovascular Health)HBQ (Health Behavior Questionnaire). The scale consists of 14 visual items with low-fat/salty and high-fat/salty food options to determine children's food consumption. Children are shown comparable foods and asked which of the two foods is more common (often).
  Trying to find out what he ate. Scale items take values of -1 for unhealthy food and +1 for healthy food. The lowest and highest scores that can be obtained from this scale are between -14 and +14. A high total score from the scale indicates that you have healthy eating habits. The internal consistency reliability coefficient of the original scale was found to be 0.76, and the test-retest reliability was 0.58 (Edmunson et al., 1996). Scale validity and reliability study for this scale was conducted by Öztürk (2010).
Parent Questionnaire | at the end of the 1th weeks
  The parent questionnaire contains 18 questions asked to parents about their children, created by the researcher by scanning the literature. The questionnaire will be scored between 18-90.

CONTACTS AND LOCATIONS:
Overall Officials: HAVVA KARADENİZ, Study Director — Research Supervisör-hkmumcu@ktu.edu.tr
Locations (1):
- Seçil Duran Yilmaz, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I may consider it in the future.